CLINICAL TRIAL: NCT03805321
Title: The Validity of Peripheral Perfusion Index to Predict Fluid Responsiveness Using Mini-fluid Challenge Test
Brief Title: The Validity of Peripheral Perfusion Index to Predict Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor of anesthesia and critical care, Cairo University
Other Study IDs: N-138-2018
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fluid therapy is an essential component of the management of patients with acute circulatory failure. Nevertheless, unnecessary administration of fluids in non-responders is harmful. Thus, the concept of fluid responsiveness has been suggested to guide fluid administration in critically ill patients to avoid either over or under-transfusion. The aim of this work is to investigate the ability of peripheral perfusion index to predict the hemodynamic response to mini-fluid challenge in patients with septic shock .

DETAILED DESCRIPTION:
The concept of fluid responsiveness has been suggested to guide fluid administration in critically ill patients to avoid either over or under-transfusion.

Several methods have been suggested to detect fluid responsiveness. Mini fluid challenge with concomitant monitoring of stroke volume is one of the most robust methods for pre-load challenge.

The main foreshortening of mini fluid challenge method is the need for a real-time cardiac output monitor, to track the instantaneous change of stroke vole with changing body position. Finding a surrogate to cardiac output to trace the effect of mini fluid challenge would make the test more applicable without the need for advanced hemodynamic monitors.

There is a growing interest in the use of perfusion indices in assessment of fluid responsiveness. Perfusion indices are measures for adequacy of oxygen delivery in peripheral tissues; thus, they were hypothesized to be possible surrogates of cardiac output. Peripheral perfusion index represents "the ratio between the pulsatile and non-pulsatile component of the light reaching the pulse oximeter" . Peripheral perfusion index has been considered as a numerical non-invasive measure for peripheral perfusion. PPI has the advantage over other perfusion indices that it a non-invasive, user-friendly monitor.

The aim of this work is to investigate the ability of peripheral perfusion index to predict the hemodynamic response to mini-fluid challenge in patients with septic shock.

Mini-fluid challenge test will be performed by infusion of 200 mL Lactated Ringer's solution over 1 minute. Velocity time integral will be monitored using Transthoracic echocardiography at the left ventricular outflow tract at the apical five-chamber view. Cardiac output will be calculated, and the patient will be considered fluid-responder if cardiac output increased by 10% after fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock patients

Exclusion Criteria:

* Evident blood loss
* Peripheral vascular disorders
* Upper limb injury or burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include septic shock patients undergoing fluid resuscitation. Patients will be enrolled during evaluation of fluid responsiveness.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Peripheral perfusion index | 2 hours
  It is a number describing the ratio between pulsatile and non-pulsatile blood flow measured by pulse oximeter. It is measured in percent. with the best value of 20% and the worst value of 0.1%

SECONDARY OUTCOMES:
Velocity time integral | 2 hours
  it is a parameter measured from Doppler across the left ventricular outflow tract. It is calculated by dividing the blood velocity by time and measured in cm
Mean arterial blood pressure | 2 hours
  Mean arterial blood pressure measured in mmHg
Central venous pressure | 2 hours
  Central venous pressure measured from a central venous catheter. It is measured in cmH2o
Systolic arterial blood pressure | 2 hours
  Systolic arterial blood pressure measured in mmHg
Diastolic arterial blood pressure | 2 hours
  Diastolic arterial blood pressure measured in mmHg
Cardiac output | 2 hours
  The amount of blood pumped by the heart in one minute. it is measured as liters per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shash, Professor, Study Director — Head of department of anesthesia, Cairo University, Egypt
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasanin A, Karam N, Mukhtar AM, Habib SF. The ability of pulse oximetry-derived peripheral perfusion index to detect fluid responsiveness in patients with septic shock. J Anesth. 2021 Apr;35(2):254-261. doi: 10.1007/s00540-021-02908-w. Epub 2021 Feb 22. PMID 33616758